CLINICAL TRIAL: NCT01397409
Title: Evaluation of AGN-150998 in Exudative Age-related Macular Degeneration (AMD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 150998-001; 2011-002526-43 (EudraCT Number); REACH Study (Other: Allergan, Inc.)
Record Dates: First submitted 2011-07-18; First posted 2011-07-19 (Estimated); Results first posted 2015-06-18 (Estimated); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Age-related Macular Degeneration
MeSH Terms: conditions — Macular Degeneration | interventions — Ranibizumab; salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (10):
- Stage 1: AGN-150998 4.2 mg (Experimental): Stage 1: AGN-150998 4.2.mg given as a single intravitreal injection.
  Interventions: Drug: AGN-150998
- Stage 1: AGN-150998 3.0 mg (Experimental): Stage 1: AGN-150998 3.0 mg given as a single intravitreal injection.
  Interventions: Drug: AGN-150998
- Stage 1: AGN-150998 2.0 mg (Experimental): Stage 1: AGN-150998 2.0 mg given as a single intravitreal injection.
  Interventions: Drug: AGN-150998
- Stage 1: AGN-150998 1.0 mg (Experimental): Stage 1: AGN-150998 1.0 mg given as a single intravitreal injection.
  Interventions: Drug: AGN-150998
- Stage 2: AGN-150998 4.2 mg (Experimental): Stage 2: AGN-150998 4,2 mg (highest tolerated dose from Stage 1) given as a single intravitreal injection at baseline. A second intravitreal injection will be given by week 16.
  Interventions: Drug: AGN-150998
- Stage 2: AGN-150998 3.0 mg (Experimental): Stage 2: AGN-150998 3.0 mg (one dose below highest tolerated dose) from Stage 1 given as a single intravitreal injection at baseline. A second intravitreal injection will be given by week 16.
  Interventions: Drug: AGN-150998
- Stage 2: ranibizumab 0.5 mg (Active Comparator): Stage 2: ranibizumab 0.5 mg given as a single intravitreal injection at baseline. A second intravitreal injection will be given by week 16.
  Interventions: Drug: ranibizumab
- Stage 3: AGN-150998 2.0 mg (Experimental): Stage 3: AGN-150998 2.0 mg given as intravitreal injections at Baseline, Weeks 4 and 8, followed by sham injections at Weeks 12 and 16.
  Interventions: Drug: AGN-150998; Other: Sham Injection
- Stage 3: AGN-150998 1.0 mg (Experimental): Stage 3: AGN-150998 1.0 mg given as intravitreal injections at Baseline, Weeks 4 and 8, followed by sham injections at Weeks 12 and 16.
  Interventions: Drug: AGN-150998; Other: Sham Injection
- Stage 3: ranibizumab 0.5 mg (Active Comparator): Stage 3: ranibizumab 0.5 mg given as intravitreal injections every 4 weeks for 16 weeks.
  Interventions: Drug: ranibizumab

INTERVENTIONS:
Drug: AGN-150998 — AGN-150998 Intravitreal injection.
  Arms: Stage 1: AGN-150998 1.0 mg; Stage 1: AGN-150998 2.0 mg; Stage 1: AGN-150998 3.0 mg; Stage 1: AGN-150998 4.2 mg; Stage 2: AGN-150998 3.0 mg; Stage 2: AGN-150998 4.2 mg; Stage 3: AGN-150998 1.0 mg; Stage 3: AGN-150998 2.0 mg
Drug: ranibizumab — Ranibizumab 0.5 mg given by intravitreal injection.
  Other Names: Lucentis®
  Arms: Stage 2: ranibizumab 0.5 mg; Stage 3: ranibizumab 0.5 mg
Other: Sham Injection — Stage 3: Sham injection at Weeks 12 and 16.
  Arms: Stage 3: AGN-150998 1.0 mg; Stage 3: AGN-150998 2.0 mg

SUMMARY:
This study is conducted in 3 stages. Stage 1 is an open-label, dose-escalation assessment of the safety of AGN-150998 administered as a single intravitreal injection to patients with advanced exudative Age-related Macular Degeneration (AMD). Stage 2 and Stage 3 are randomized, double-masked, comparisons of the safety and treatment effects on retinal edema and best-corrected visual acuity (BCVA) of AGN-150998 and ranibizumab in treatment-naive patients with exudative AMD. Study medication is administered as needed in Stage 2 and with a fixed-dosing schedule in Stage 3. The study objectives are (1) to identify the highest tolerated dose of AGN-150998, (2) to assess the safety and duration of treatment effects on retinal edema and BCVA, and (3) to characterize the systemic pharmacokinetic profile of AGN-150998.

ELIGIBILITY:
Inclusion Criteria:

* Exudative age-related macular degeneration
* Best-corrected visual acuity between 20/32 and 20/320 in the study eye

Exclusion Criteria:

* Near-sightedness of 8 diopters or more
* Uncontrolled glaucoma in the study eye
* Cataract surgery or Lasik within the last 3 months
* Any active ocular infection or inflammation

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 271 (Actual)
Dates: Start 2011-09-01 (Actual); Primary Completion 2014-03-31 (Actual); Study Completion 2014-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (8):
- Phoenix, Arizona, United States
- Sydney, New South Wales, Australia
- Vienna, Austria
- Créteil, France
- Bonn, Germany
- Tel Aviv, Israel
- Florence, Italy
- Binningen, Switzerland

REFERENCES:
- [Background] Callanan D, Kunimoto D, Maturi RK, Patel SS, Staurenghi G, Wolf S, Cheetham JK, Hohman TC, Kim K, Lopez FJ, Schneider S. Double-Masked, Randomized, Phase 2 Evaluation of Abicipar Pegol (an Anti-VEGF DARPin Therapeutic) in Neovascular Age-Related Macular Degeneration. J Ocul Pharmacol Ther. 2018 Dec;34(10):700-709. doi: 10.1089/jop.2018.0062. Epub 2018 Nov 9. PMID 30412448

RESULTS

PARTICIPANT FLOW:
Groups:
- Stage 1: AGN-150998 4.2 mg: Stage 1: AGN-150998 4.2 mg given as a single intravitreal injection.
- Stage 2: AGN-150998 4.2 mg: Stage 2: AGN-150998 4.2 mg (highest tolerated dose from Stage 1) given as a single intravitreal injection at baseline. A second intravitreal injection will be given by week 16.
- Stage 2: AGN-150998 3.0 mg: Stage 2: AGN-150998 3.0 mg (one dose below highest tolerated dose from Stage 1) given as a single intravitreal injection at baseline. A second intravitreal injection will be given by week 16.
Period: Stage 1
Arm/Group | Stage 1: AGN-150998 4.2 mg | Stage 1: AGN-150998 3.0 mg | Stage 1: AGN-150998 2.0 mg | Stage 1: AGN-150998 1.0 mg | Stage 2: AGN-150998 4.2 mg | Stage 2: AGN-150998 3.0 mg | Stage 2: Ranibizumab 0.5 mg | Stage 3: AGN-150998 2.0 mg | Stage 3: AGN-150998 1.0 mg | Stage 3: Ranibizumab 0.5 mg
Started | 9 | 6 | 6 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 9 | 6 | 6 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Stage 2
Arm/Group | Stage 1: AGN-150998 4.2 mg | Stage 1: AGN-150998 3.0 mg | Stage 1: AGN-150998 2.0 mg | Stage 1: AGN-150998 1.0 mg | Stage 2: AGN-150998 4.2 mg | Stage 2: AGN-150998 3.0 mg | Stage 2: Ranibizumab 0.5 mg | Stage 3: AGN-150998 2.0 mg | Stage 3: AGN-150998 1.0 mg | Stage 3: Ranibizumab 0.5 mg
Started | 0 | 0 | 0 | 0 | 67 | 58 | 58 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 59 | 54 | 58 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 8 | 4 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 6 | 3 | 0 | 0 | 0 | 0
Not completed — Personal Reasons | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Other Miscellaneous Reasons | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Period: Stage 3
Arm/Group | Stage 1: AGN-150998 4.2 mg | Stage 1: AGN-150998 3.0 mg | Stage 1: AGN-150998 2.0 mg | Stage 1: AGN-150998 1.0 mg | Stage 2: AGN-150998 4.2 mg | Stage 2: AGN-150998 3.0 mg | Stage 2: Ranibizumab 0.5 mg | Stage 3: AGN-150998 2.0 mg | Stage 3: AGN-150998 1.0 mg | Stage 3: Ranibizumab 0.5 mg
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 23 | 25 | 16
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 21 | 25 | 16
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Other Miscellaneous Reasons | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Stage 1: AGN-150998 4.2 mg | Stage 1: AGN-150998 3.0 mg | Stage 1: AGN-150998 2.0 mg | Stage 1: AGN-150998 1.0 mg | Stage 2: AGN-150998 4.2 mg | Stage 2: AGN-150998 3.0 mg | Stage 2: Ranibizumab 0.5 mg | Stage 3: AGN-150998 2.0 mg | Stage 3: AGN-150998 1.0 mg | Stage 3: Ranibizumab 0.5 mg | Total
Number analyzed (Participants) | 9 | 6 | 6 | 3 | 67 | 58 | 58 | 23 | 25 | 16 | 271
Age, Continuous [Mean (Full Range); unit: Years] | 82.3 [68 to 89] | 75.3 [62 to 86] | 79.3 [72 to 91] | 67.7 [64 to 71] | 80.4 [58 to 95] | 78.6 [63 to 94] | 78.5 [59 to 92] | 77.9 [67 to 89] | 75.5 [54 to 91] | 76.5 [53 to 86] | 77.2 [53 to 95]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 2 | 4 | 2 | 34 | 35 | 38 | 13 | 18 | 8 | 159
  Male | 4 | 4 | 2 | 1 | 33 | 23 | 20 | 10 | 7 | 8 | 112

OUTCOME MEASURES:

1. Primary Outcome: Highest Tolerated Dose (HTD) of AGN-150998
Description: Stage 1 evaluated the safety of a single intravitreal injection of AGN-150998 with doses ranging from 1.0 to 4.2 mg.
Time Frame: 24 Weeks
Population: Safety population included all treated participants.
Measure: Number; unit: mg
Groups:
- Stage 1 All Participants: Participants in Stage 1 received an intravitreal injection of AGN-150998 with doses ranging from 1.0 to 4.2 mg.
Arm/Group | Stage 1 All Participants
Number analyzed (Participants) | 24
mg | 4.2

2. Primary Outcome: Stage 1: Change From Baseline in Central Retinal Thickness (CRT) in the Study Eye
Description: CRT was assessed using spectral domain optical coherence tomography (SD-OCT), a non-invasive diagnostic system providing high-resolution imaging sections of the retina. SD-OCT was performed in the study eye after pupil dilation. A negative change from Baseline indicated improvement.
Time Frame: Baseline, Week 4
Population: Safety population included all treated participants.
Measure: Mean (Standard Deviation); unit: microns
Arm/Group | Stage 1: AGN-150998 4.2 mg | Stage 1: AGN-150998 3.0 mg | Stage 1: AGN-150998 2.0 mg | Stage 1: AGN-150998 1.0 mg
Number analyzed (Participants) | 9 | 6 | 6 | 3
microns
  Baseline | 527.6 (126.79) | 540.3 (284.34) | 500.3 (155.65) | 564.3 (115.68)
  Change from Baseline at Week 4 (n=9,6,6,2) | -185.4 (161.23) | -239.5 (234.03) | -212.3 (182.94) | -113.5 (135.06)

3. Primary Outcome: Stage 2: Time Between Baseline Treatment and Recurrence of Active Disease
Description: Recurrence of Active Disease was based on Best Corrected Visual Acuity (BCVA), Central Retinal Thickness (CRT) values as evaluated by the Central Reading Center (CRC) and the investigator assessments of haemorrhage.
Time Frame: Baseline, Week 16
Population: Per-protocol Population included all treated participants who received all scheduled treatments.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Stage 2: AGN-150998 4.2 mg | Stage 2: AGN-150998 3.0 mg | Stage 2: Ranibizumab 0.5 mg
Number analyzed (Participants) | 65 | 57 | 57
days | 59.0 [43.0 to 109.0] | 57.0 [43.0 to 86.0] | 57.0 [43.0 to 85.0]

4. Primary Outcome: Stage 3: Change From Baseline in Best Corrected Visual Acuity (BCVA) in the Study Eye
Description: BCVA is measured using an eye chart and is reported as the number of letters read correctly (ranging from 0 to 100 letters) in the study eye. The lower the number of letters read correctly on the eye chart, the worse the vision (or visual acuity). An increase in the number of letters read correctly means that vision has improved.
Time Frame: Baseline, Week 16
Population: Modified-Intent-to-Treat (mITT) Population
Measure: Mean (Standard Deviation); unit: letters
Arm/Group | Stage 3: AGN-150998 2.0 mg | Stage 3: AGN-150998 1.0 mg | Stage 3: Ranibizumab 0.5 mg
Number analyzed (Participants) | 23 | 25 | 16
letters
  Baseline | 58.5 (14.29) | 58.4 (13.49) | 60.4 (16.41)
  Change from Baseline at Week 16 | 8.2 (7.89) | 6.3 (7.81) | 5.3 (11.08)

5. Secondary Outcome: Stage 2: Time Between Second Treatment and Recurrence of Active Disease
Description: Recurrence of active disease is defined as the time in days to escape to standard of care. Time is calculated as (date of Escaping to Standard of Care/Censoring minus the date of the Second Injection) +1.
Time Frame: 32 Weeks
Population: mITT Population
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Stage 2: AGN-150998 4.2 mg | Stage 2: AGN-150998 3.0 mg | Stage 2: Ranibizumab 0.5 mg
Number analyzed (Participants) | 62 | 55 | 58
days | 85.0 [57.0 to 118.0] | 112.0 [60.0 to NA] — 75% Upper Limit not estimated. | 111.0 [57.0 to NA] — 75% Upper Limit not estimated.

6. Secondary Outcome: Stage 2: Change From Baseline in Central Retinal Thickness (CRT) in the Study Eye
Description: as for outcome 2
Time Frame: Baseline, Week 4
Population: Per-protocol Population included all treated participants who received all scheduled treatments.
Measure: Mean (Standard Deviation); unit: microns
Arm/Group | Stage 2: AGN-150998 4.2 mg | Stage 2: AGN-150998 3.0 mg | Stage 2: Ranibizumab 0.5 mg
Number analyzed (Participants) | 65 | 57 | 57
microns
  Baseline | 524.6 (170.71) | 507.3 (139.88) | 497.1 (122.04)
  Change from Baseline at Week 4 (n=61,56,57) | -179.5 (123.76) | -155.3 (109.13) | -157.3 (121.95)

7. Secondary Outcome: Stage 2: Change From Baseline in Best Corrected Visual Acuity (BCVA) in the Study Eye
Description: as for outcome 4
Time Frame: Baseline, Week 4
Population: Per-protocol Population included all treated participants who received all scheduled treatments.
Measure: Mean (Standard Deviation); unit: letters
Arm/Group | Stage 2: AGN-150998 4.2 mg | Stage 2: AGN-150998 3.0 mg | Stage 2: Ranibizumab 0.5 mg
Number analyzed (Participants) | 65 | 57 | 57
letters
  Baseline | 54.5 (13.90) | 52.7 (12.62) | 55.4 (13.00)
  Change from Baseline at Week 4 (n=62,56,57) | 4.7 (9.71) | 8.4 (11.51) | 5.9 (64.0)

8. Secondary Outcome: Stage 3: Change From Baseline in Central Retinal Thickness (CRT) in the Study Eye
Description: as for outcome 2
Time Frame: Baseline, Week 4
Population: Per-protocol Population included all treated participants who received all scheduled treatments.
Measure: Mean (Standard Deviation); unit: microns
Arm/Group | Stage 3: AGN-150998 2.0 mg | Stage 3: AGN-150998 1.0 mg | Stage 3: Ranibizumab 0.5 mg
Number analyzed (Participants) | 23 | 25 | 16
microns
  Baseline | 466.0 (125.96) | 526.1 (165.09) | 463.3 (94.56)
  Change from Baseline at Week 4 | -119.8 (68.50) | -168.3 (137.07) | -98.4 (65.22)

9. Secondary Outcome: Stage 3: Change From Baseline in BCVA in the Study Eye
Description: as for outcome 4
Time Frame: Baseline, Week 4
Population: Per-protocol Population included all treated participants who received all scheduled treatments.
Measure: Mean (Standard Deviation); unit: letters
Arm/Group | Stage 3: AGN-150998 2.0 mg | Stage 3: AGN-150998 1.0 mg | Stage 3: Ranibizumab 0.5 mg
Number analyzed (Participants) | 23 | 25 | 16
letters
  Baseline | 58.5 (14.29) | 58.4 (13.49) | 60.4 (16.41)
  Change from Baseline at Week 4 | 5.0 (7.40) | 4.6 (5.98) | 3.9 (6.01)

ADVERSE EVENTS:
Arm/Group | Stage 1: AGN-150998 4.2 mg | Stage 1: AGN-150998 3.0 mg | Stage 1: AGN-150998 2.0 mg | Stage 1: AGN-150998 1.0 mg | Stage 2: AGN-150998 4.2 mg | Stage 2: AGN-150998 3.0 mg | Stage 2: Ranibizumab 0.5 mg | Stage 3: AGN-150998 2.0 mg | Stage 3: AGN-150998 1.0 mg | Stage 3: Ranibizumab 0.5 mg
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/6 | 1/6 | 0/3 | 11/67 | 6/58 | 5/58 | 0/23 | 0/25 | 0/16
Other Adverse Events (participants affected / at risk) | 3/9 | 5/6 | 4/6 | 2/3 | 51/67 | 35/58 | 35/58 | 10/23 | 15/25 | 9/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Stage 1: AGN-150998 4.2 mg (N=9) | Stage 1: AGN-150998 3.0 mg (N=6) | Stage 1: AGN-150998 2.0 mg (N=6) | Stage 1: AGN-150998 1.0 mg (N=3) | Stage 2: AGN-150998 4.2 mg (N=67) | Stage 2: AGN-150998 3.0 mg (N=58) | Stage 2: Ranibizumab 0.5 mg (N=58) | Stage 3: AGN-150998 2.0 mg (N=23) | Stage 3: AGN-150998 1.0 mg (N=25) | Stage 3: Ranibizumab 0.5 mg (N=16)
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Uveitus (Eye disorders) | 0 | 0 | 0 | 0 | 3 | 2 | 0 | 0 | 0 | 0
Anterior chamber inflammation (Eye disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Vitritis (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Aortic valve stenosis (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Choroiditis (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Endophthalmitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Glaucoma (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Optic ischaemic neuropathy (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Retinal artery occlusion (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Temporal arteritis (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Atypical pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Stage 1: AGN-150998 4.2 mg (N=9) | Stage 1: AGN-150998 3.0 mg (N=6) | Stage 1: AGN-150998 2.0 mg (N=6) | Stage 1: AGN-150998 1.0 mg (N=3) | Stage 2: AGN-150998 4.2 mg (N=67) | Stage 2: AGN-150998 3.0 mg (N=58) | Stage 2: Ranibizumab 0.5 mg (N=58) | Stage 3: AGN-150998 2.0 mg (N=23) | Stage 3: AGN-150998 1.0 mg (N=25) | Stage 3: Ranibizumab 0.5 mg (N=16)
Palpitations (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ventricular extrasystoles (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anterior chamber inflammation (Eye disorders) | 1 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0
Retinal pigment epithelial tear (Eye disorders) | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 0
Conjunctival haemorrhage (Eye disorders) | 0 | 1 | 1 | 1 | 9 | 3 | 5 | 1 | 2 | 0
Eye irritation (Eye disorders) | 0 | 1 | 1 | 0 | 5 | 2 | 2 | 1 | 1 | 0
Anterior chamber cell (Eye disorders) | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Anterior chamber flare (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eye pain (Eye disorders) | 0 | 1 | 0 | 0 | 6 | 3 | 4 | 2 | 1 | 1
Hyalosis asteroid (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Macular oedema (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Foreign body sensation in eyes (Eye disorders) | 0 | 0 | 1 | 0 | 4 | 0 | 1 | 0 | 1 | 1
Retinal haemorrhage (Eye disorders) | 0 | 0 | 0 | 1 | 6 | 3 | 4 | 0 | 3 | 2
Urinary tract infection (Infections and infestations) | 1 | 1 | 0 | 0 | 1 | 0 | 2 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0 | 0 | 0 | 4 | 2 | 1 | 0 | 0 | 1
Viral upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vitreous detachment (Eye disorders) | 0 | 0 | 0 | 0 | 5 | 6 | 2 | 2 | 2 | 0
Visual acuity reduced (Eye disorders) | 0 | 0 | 0 | 0 | 5 | 3 | 3 | 0 | 0 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vitritis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 1 | 0
Vitreous floaters (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 1 | 3 | 1
Dry eye (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 4 | 2 | 2 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 3 | 1 | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 3 | 3 | 1 | 0 | 1
Age-related macular degeneration (Eye disorders) | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 1 | 1
Macular scar (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Choroidal neovascularisation (Eye disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 0 | 0 | 1
Eye pruritus (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1
Ocular discomfort (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1
Visual impairment (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 1 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.